CLINICAL TRIAL: NCT04085666
Title: A Phase 1, Multi-center, Randomized, Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Pharmacodynamics, Safety, Tolerability and Pharmacokinetics of a Single Oral Dose of CDX-6114 in Patients With Phenylketonuria (PKU).
Brief Title: Pharmacodynamics, Safety, Tolerability and Pharmacokinetics of CDX-6114 in Patients With Phenylketonuria (PKU)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CDX6114-002
Record Dates: First submitted 2019-08-03; First posted 2019-09-11 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st Confinement Period in Unit (Experimental): Randomized to treatment with either CDX-6114 or matching Placebo
  Interventions: Drug: CDX 6114; Other: Matching Placebo
- 2nd Confinement Period in Unit (Experimental): Randomized to treatment with either CDX-6114 or matching Placebo
  Interventions: Drug: CDX 6114; Other: Matching Placebo

INTERVENTIONS:
Drug: CDX 6114 — CDX-6114 for oral administration is formulated in phosphate buffer, which also includes mannitol and poloxamer.The vehicle solution provided is identical to the CDX-6114 oral solution except for the active drug.
Other: Matching Placebo — The placebo oral dosing solution will also be supplied as an approximately 240 mL oral solution and will be made up of the phosphate buffer diluent and the caramel flavoring.

SUMMARY:
This study is an international, multi-center, randomized, double-blind, placebo-controlled, two-treatment, two-period cross-over study to evaluate the pharmacodynamics, safety, tolerability and pharmacokinetics of a single oral dose of CDX-6114 in patients with phenylketonuria (PKU).

ELIGIBILITY:
* Inclusion criteria

  1. Male and female patients between the ages of 18 and 55 years (inclusive) with a diagnosis of classical PKU by either a historical blood Phe concentration of > 1200 mol/L at any time or a genetic diagnosis of PKU.
  2. Patients capable of following dietary instructions to maintain protein intake stable throughout the study duration based on principal investigator and dietician assessment.
  3. Patients with a blood Phe concentration < 1200mol/L at screening.
  4. Have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
  5. Patients must be in good general health, as determined by the PI or delegate, based on a medical evaluation including detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG) and clinical laboratory tests.
  6. Male patients (unless surgically sterilised) and their female spouse/partner(s) who are of childbearing potential:

     1. Must agree to stay abstinent (where abstinence is the preferred and usual life-style of the patient), starting at screening and continuing throughout the clinical study period, and for 90 days after last study drug administration.

        Or
     2. Must be using highly effective contraception starting at screening and continuing throughout the clinical study period, and for 90 days after last study drug administration. Highly effective contraception is defined as follows:

     i. Injectable or implantable hormones ii. Intrauterine device iii. Surgical sterilisation iv. Sterilisation implant device v. Combined oral contraceptives vi. Use of a condom plus oral or injectable or implantable or intrauterine contraception

     c. These requirements do not apply to participants in a same sex relationship.
  7. Male patients must agree not to donate sperm starting at screening and continuing throughout the clinical study period, and for 90 days after last study drug administration.
  8. Female patients of childbearing potential and their spouse/partner(s):

     1. Must agree not to become pregnant during the clinical study period and for 30 days after last study drug administration.
     2. Must have a negative serum pregnancy test at screening.
     3. If heterosexually active, must agree to consistently use a form of highly effective contraception, starting at screening and continuing throughout the clinical study period, and for 30 days after last study drug administration. Highly effective contraception is defined as follows:

     i. Injectable or implantable hormones ii. Intrauterine device iii. Surgical sterilisation iv. Sterilisation implant device v. Surgical sterilisation of the male partner vi. Combined oral contraceptives vii. Use of a condom plus oral or injectable or implantable or intrauterine contraception

     Or

     d. Must agree to stay abstinent (where abstinence is the preferred and usual life-style of the patient), starting at screening and continuing throughout the clinical study period, and for 30 days after last study drug administration.

     e. These requirements do not apply to participants in a same sex relationship.
  9. Female patients of non-childbearing potential:

     1. Must have a confirmed clinical history of sterility (e.g. the patient is without a uterus).

        Or
     2. Must be postmenopausal as defined as amenorrhea for at least 1 year prior to screening and a laboratory confirmed serum follicle stimulating hormone (FSH) level ≥ 40mIU/mL or similar value considered to be in the menopausal range.
  10. Female patients must agree not to breastfeed from screening, throughout the clinical study period, and until 90 days after last study drug administration.
  11. Female patients must agree not to donate ova from screening, throughout the clinical study period, and until 90 days after last study drug administration.
  12. Patient must be competent to understand the nature of the study and capable of giving written informed consent. Be willing to report for the scheduled study visits and communicate to study personnel about adverse events and concomitant medication use.
  13. Patient agrees not to participate in another interventional study while participating in the present clinical study.

Exclusion criteria

1. Female patient who has been pregnant within the 6 months prior to screening or breastfeeding within the 3 months prior to screening.
2. Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies and childhood asthma) at time of screening.
3. Current or chronic history of gastrointestinal illness or conditions interfering with normal gastrointestinal anatomy or motility. Examples include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, irritable bowel syndrome (IBS) or celiac sprue.
4. Evidence or history of gastrointestinal symptoms that could lead to the assumption of an underlying gastrointestinal impairment.
5. Treatment with any anti-platelet and/or anticoagulant medication.
6. Evidence or history of specific food intolerance. Examples include coeliac disease, severe lactose or dairy food intolerance or a severe intolerance to any food/ingredient included in the standard breakfast.
7. Any positive result, on screening, for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCV) or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2).
8. A positive drug/alcohol result.
9. Patient has a history of exceeding > 21 units of alcohol/week for male patients or > 14 units of alcohol/week for female patients within the 3 months prior to screening. One unit of alcohol is equivalent to 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits.
10. Patient has a history of regular smoking (daily or most days in a week) or the use of nicotine products (3 or more nicotine-containing products) who would be unable to abstain from smoking during the confinement periods in the Phase 1 Unit.
11. Patient has used any recreational drugs of abuse within the 3 months prior to screening.
12. Patient has a pulse rate ≤ 50 or ≥ 100 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg at screening (excluding white-coat hypertension; therefore, a repeat test showing results within range will be acceptable).
13. Patient has any clinically significant abnormalities at screening in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the PI or delegate, which may interfere with the interpretation of QTc interval changes including abnormal ST-T wave morphology.
14. Patient has prolonged QTcF (QT interval corrected for heart rate using Fridericia's formula) > 450 ms for male patients or > 470 ms for female patients, or a shortened QTcF < 300 ms or a family history of prolonged QT syndrome, at screening.
15. Patient has any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis at screening as judged by the PI or delegate, including: Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT) or Total bilirubin (TBL) more than 2.0 times above the Upper Limit of Normal (ULN).
16. Plasma donation within the 14 days prior to screening or any whole blood donation/significant blood loss > 500 mL during the 3 months prior to screening.
17. Treatment with any Investigational Drug or Device/Treatment within the 30 days prior to the first administration of study drug.
18. Use of any prescribed or non-prescribed medication including herbal medicines, antacids and analgesics (other than anti-hypertensive drugs, oral contraceptives, paracetamol or multi-vitamins) for the two weeks prior to the initial administration of the study medication or up to a minimum of 5 times the half-life of the medication if it has a long half-life.
19. Known allergy or adverse reaction history to any of the oral dose formulation components e.g. mannitol.
20. Use of Sapropterin (KUVAN) or pegylated phenylalanine ammonia lyase (Palinzyk) or SYNB1618 or any Phenylalanine-lowering drug within the last 4 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in concentration of post parandial plasma level of Phe will be summarized over time for each treatment | Within 30 minutes, within 10 minutes and immediately prior to dosing, and then at 15 minutes, 30 minutes, 1hours, 1.5, 2,4 and 5hours after dosing on both Day 1 and Day 8
  Blood samples will be collected at the following time points to determine the postprandial plasma levels of Phe following single does of CDX-6114
Change in concentration of post parandial plasma level of CA will be summarized over time for each treatment | Within 30 minutes, within 10 minutes and immediately prior to dosing, and then at 15 minutes, 30 minutes, 1hours, 1.5, 2,4 and 5hours after dosing on both Day 1 and Day 8
  Blood samples will be collected at the following time points to determine the postprandial plasma levels of CA following single does of CDX-6114
Change in the peak Phe concentration in Plasma will be summarized by treatment | Within 30 minutes, within 10 minutesand immediately prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8
  Blood samples will be collected at the following time points to determine the Peak Phe plasma concentration follwoing a single, oral dose of CDX-6114
Change in the peak CA concentration in Plasma will be summarized by treatment | Within 30 minutes, within 10 minutesand immediately prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8
  Blood samples will be collected at the following time points to determine the Peak CA plasma concentration following a single, oral dose of CDX-6114
Phe Area under the plasma concentration versus time curve (AUC) , over a 5-hour period, following dosing and the standardized breakfast | Within 30 minutes, within 10 minutesand immediately prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8
  Blood samples will be collected at the following time points to determine the Phe AUC following a single, oral dose of CDX-6114
CA Area under the plasma concentration versus time curve (AUC) , over a 5-hour period, following dosing and the standardized breakfast | Within 30 minutes, within 10 minutesand immediately prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8
  Blood samples will be collected at the following time points to determine the CA AUC following a single, oral dose of CDX-6114

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) will be measured | Within 30 minutes, within 10 minutes and immediately prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by Adverse events monitoring
The serum levels of CDX-6114 will be summarized descriptively over time | Within 30 minutes, within 10 minutes and immediately prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8
  Blood will be collected for pharmacokinetic analysis of CDX-6114 at the following time points follwoing a single oral dose of CDX-6114
Absolute values and changes from baseline in blood pressure measurements will be summarized over time for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by blood pressure monitoring
Absolute values and changes from baseline in Heart rate measurements will be summarized over time for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by Heart rate monitoring
Absolute values and changes from baseline in Respiratory rate measurements will be summarized over time for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by Respiratory rate monitoring
Absolute values and changes from baseline in body temperature (in Fahrenheit or Celsius) measurements will be summarized over time for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by Body temperature monitoring
Absolute values and changes from baseline in 12 lead Electrocardiogram (ECG) measurements will be summarized over time for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by 12 lead ECG including P Wave, QRS Complex, QT Interval
Absolute values of Weight measurements will be summarized over time for each treatment using a weighing scale in Kg or pounds | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1hr, 1.5hr, 2hr, 4hr and 5hr after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by weight monitoring
Absolute blood composition values and changes from baseline to the last post-dose time-point will be summarized for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by laboratory assessments as Haematology and Coagulation
Absolute urine composition values and changes from baseline to the last post-dose time-point will be summarized for each treatment | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1, 1.5, 2, 4 and 5hours after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by routine urinalysis laboratory assessments
Assesment of the incidence of Treatment-Emergent Antibodies | Assesments will be done on day 1 and day 8. Blood will be collected for analysis within 30 minutes prior to dosing on Day 1 and Day 8 and again at the End of Study Visit ( through study completion , an avearge of 8 to 10 weeks)
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by assessment for development of anti-CDX-6114 antibodies
absolute values of height measurements will be summarized over time for each treatment using length measurement scale in centimeters or inches | Within 30 minutes prior to dosing, and then at 15 minutes, 30 minutes, 1hr, 1.5hr, 2hr, 4hr and 5hr after dosing on both Day 1 and Day 8.
  The safety and tolerability of CDX-6114 following single dose oral administration assesed by height examination using Lenght scale

CONTACTS AND LOCATIONS:
Overall Officials: Damon Bell, Principal Investigator — Linear Clinical Research; Tim Heise, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (2):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany